CLINICAL TRIAL: NCT01480635
Title: Evaluation of the PillCam Colon Capsule Endoscopy (PCCE) After Incomplete Colonoscopy
Brief Title: PillCam Colon 2 Capsule Endoscopy (PCCE) After Incomplete Colonoscopy
Acronym: PCCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bethesda Krankenhaus (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: PV3467
Record Dates: First submitted 2011-10-13; First posted 2011-11-29 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-10

CONDITIONS: Colonoscopy
Keywords: Incomplete Colonoscopy; Efficacy of PillCam Colon2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Incomplete Colonoscopy

SUMMARY:
Purpose of study:

To evaluate the efficacy of PillCam Colon2 in subjects with an incomplete standard colonoscopy

Study design: 4 centers, prospective, cohort study Number of subjects: 74 subjects

Subject population: Patients that are indicated for colonoscopy, who are suspected or known to suffer from colonic diseases and had an incomplete standard colonoscopy

Control group: None Procedure Duration: Approximately 10-12 hours Duration of Follow up: One week follow up Duration of study: 12 months

Primary objectives: Evaluation of the efficacy of PillCam Colon2 to visualize the colon segment not reached by an incomplete standard colonoscopy Evaluation of distribution of excretion of capsules over time

ELIGIBILITY:
Inclusion Criteria:

* Subject is >/= 18 years
* Subject is suspected/known to suffer from large bowel disease and was clinically referred for colonoscopy.
* Standard colonoscopy could not be performed completely in spite of adequate bowel cleansing and in the absence of a relevant colonic or rectal stenosis. Reasons for incomplete colonoscopy: adhesions, elongated colon, repeatedly forming loops, difficult procedure(time to reach the cecum >45 min), adverse reaction to sedation requiring termination of colonoscopy

Exclusion Criteria:

* Subject has dysphagia or any swallowing disorder
* Subject has severe congestive heart failure or renal insufficiency
* Subject with high risk for capsule retention
* Subject has a cardiac pacemakers or other implanted electromedical devices
* Subject has any allergy or other contraindication to the medications used in the study
* Subject is expected to undergo MRI examination 7 days after capsule ingestion Subject has any condition, which precludes compliance with study and/or device instructions.
* Women who are pregnant or nursing at the time of screening and/or during the study period, or are of child bearing potential without medically acceptable methods of contraception
* Subject suffers from life threatening conditions
* Subject currently participating in another clinical study
* Colonoscopy had been performed by a physician who has experience of <1000 complete colonoscopies
* Exchange of the endoscope had been performed because complete colonoscopy was impossible with the standard endoscope
* Time interval between incomplete colonoscopy and capsule endoscopy >30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are indicated for colonoscopy, who are suspected or known to suffer from colonic diseases and had an incomplete standard colonoscopy
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-07 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of PillCam Colon2 to visualize the colon segment not reached by an incomplete standard colonoscopy | One week follow up
  Study endpoint: Number of patients in whom capsule colonoscopy visualizes the complete segments missed by prior incomplete standard colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Keuchel, Dr., Principal Investigator — Bethesda Krankenhaus Bergedorf, Hamburg, Germany
Locations (6):
- Germany (6):
  - Bethesda Krankenhaus Bergedorf, Hamburg, Hamburg
  - Asklepios Klinik Altona, Hamburg, Hamburg
  - Ev. Krankenhaus Düsseldorf, Düsseldorf
  - Gastroenterologische Praxis, Düsseldorf
  - Klinikum der J.W. Goethe-Universität, Medizinische Klinik 1, Frankfurt
  - Klinikum der Stadt Ludwigshafen am Rhein, Ludwigshafen